CLINICAL TRIAL: NCT03375190
Title: A Comparison of Peripheral Nerve Catheter Securement Techniques at the Insertion Site in Healthy Volunteers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Pro00081185
Record Dates: First submitted 2017-12-05; First posted 2017-12-15 (Actual); Last update posted 2018-05-14 (Actual); Status verified 2018-05

CONDITIONS: Regional Anesthesia Morbidity
MeSH Terms: interventions — Bandages; Adhesives; Benzoin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Dressing (Experimental): Transparent film dressing (TegadermTM CHG Chlorhexidine Gluconate IV Securement Dressing, 3M Health Care, St. Paul, MN, USA) alone
  Interventions: Other: Dressing
- Dressing + adhesive (Experimental): Transparent film dressing + topical skin adhesive (SwiftSetTM Topical Skin Adhesive, CovidienTM, Devon, UK) at insertion site
  Interventions: Other: Dressing + adhesive
- Dressing + adhesive + strips (parallel) (Experimental): Transparent film dressing + topical skin adhesive + reinforced skin closure strips (Steri-StripTM, 3M Health Care, St. Paul, MN, USA) placed parallel to long axis of catheter
  Interventions: Other: Experimental: Dressing + adhesive + strips (parallel)
- Dressing + adhesive + strips (perpend) (Experimental): Transparent film dressing + topical skin adhesive + reinforced skin closure strips (Steri-StripTM, 3M Health Care, St. Paul, MN, USA) placed perpendicular to long axis of catheter
  Interventions: Other: Experimental: Dressing + adhesive + strips (perpend)
- Dressing + adhesive + strips + benzoin (Experimental): Transparent film dressing + topical skin adhesive + skin closure strips + topical benzoin (Compound Tincture of Benzoin USP 10%, Professional Disposables International, Inc., Orangeburg, NY, USA) spread in a 12 centimeter by 14 centimeter area around the insertion site
  Interventions: Other: Experimental: Dressing + adhesive + strips + benzoin
- Dressing + adhesive + strips + spray (Experimental): Transparent film dressing + topical skin adhesive + skin closure strips + medical adhesive spray (AdaptTM Medical Adhesive, Hollister Incorporated, Libertyville, IL, USA) in a 12 centimeter by 14 centimeter area around the insertion site
  Interventions: Other: Experimental: Dressing + adhesive + strips + spray

INTERVENTIONS:
Other: Dressing — Transparent film dressing (TegadermTM CHG Chlorhexidine Gluconate IV Securement Dressing, 3M Health Care, St. Paul, MN, USA) alone
  Arms: Dressing
Other: Dressing + adhesive — Transparent film dressing + topical skin adhesive (SwiftSetTM Topical Skin Adhesive, CovidienTM Devon, UK) at insertion site
  Arms: Dressing + adhesive
Other: Experimental: Dressing + adhesive + strips (parallel) — Transparent film dressing + topical skin adhesive + reinforced skin closure strips (Steri-StripTM, 3M Health Care, St. Paul, MN, USA) placed parallel to long axis of catheter
  Arms: Dressing + adhesive + strips (parallel)
Other: Experimental: Dressing + adhesive + strips (perpend) — Transparent film dressing + topical skin adhesive + reinforced skin closure strips (Steri-StripTM, 3M Health Care, St. Paul, MN, USA) placed perpendicular to long axis of catheter
  Arms: Dressing + adhesive + strips (perpend)
Other: Experimental: Dressing + adhesive + strips + benzoin — Transparent film dressing + topical skin adhesive + skin closure strips + topical benzoin (Compound Tincture of Benzoin USP 10%, Professional Disposables International, Inc., Orangeburg, NY, USA) spread in a 12 centimeter by 14 centimeter area around the insertion site
  Arms: Dressing + adhesive + strips + benzoin
Other: Experimental: Dressing + adhesive + strips + spray — Transparent film dressing + topical skin adhesive + skin closure strips + medical adhesive spray (AdaptTM Medical Adhesive, Hollister Incorporated, Libertyville, IL, USA) in a 12 centimeter by 14 centimeter area around the insertion site
  Arms: Dressing + adhesive + strips + spray

SUMMARY:
Continuous peripheral nerve block catheters are used for prolonged analgesia, but are often associated with complications such as catheter failure or dislodgement. This is a single center, prospective study to compare peripheral nerve catheter securement techniques at the insertion site in healthy volunteers.

DETAILED DESCRIPTION:
This study will involve the placement of subcutaneous peripheral nerve catheters in healthy volunteers utilizing 6 different securement techniques. The primary outcome is the force required to dislodge the peripheral nerve catheter by 1 centimeter as measured by a dynamometer in Newtons. The secondary endpoint will be the force required to disrupt the catheter dressing.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-85 years
* American Society of Anesthesiologists Physical Status I-II
* BMI 18-30 kg/m2

Exclusion Criteria:

* Inability to cooperate with or understand protocol
* Inability to understand or speak English
* Allergy to adhesive or tape
* Local infection in lower extremities
* Neurologic deficit or disorder
* Anticoagulation

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2018-02-15 (Actual); Primary Completion 2018-02-28 (Actual); Study Completion 2018-02-28 (Actual)

PRIMARY OUTCOMES:
Force required to dislodge catheter by 1 centimeter | 1 study day
  This force will be measured using a dynamometer in Newtons

SECONDARY OUTCOMES:
Force required to disrupt catheter dressing | 1 study day
  This force will be measured using a dynamometer in Newtons

CONTACTS AND LOCATIONS:
Overall Officials: Michael Shaughnessy, MD, Principal Investigator — Duke UMC
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kumar AH, MacLeod DB, Kumar KR, Ray N, Gadsden J. Comparison of perineural catheter fixation methods: a volunteer study. Anaesthesia. 2021 May;76(5):714-716. doi: 10.1111/anae.15372. Epub 2021 Jan 6. No abstract available. PMID 33406276